CLINICAL TRIAL: NCT00001230
Title: Host Response to Infection and Treatment in the Filarial Diseases of Humans
Brief Title: Host Response to Infection and Treatment in Filarial Diseases
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 880083; 88-I-0083
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-28 (Actual); Status verified 2026-01-26

CONDITIONS: Filariasis; Helminthiasis; Parasitic Infection; Mansonelliasis; Onchocerciasis
Keywords: Wuchereria Bancrofti; Loa Loa; Brugia Malayi; Onchocerca Volvulus; Filarial Infection; Natural History
MeSH Terms: conditions — Filariasis; Helminthiasis; Parasitic Diseases; Mansonelliasis; Onchocerciasis | interventions — Diethylcarbamazine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Patients that have, or are suspected of having, one of the filarial infections affecting humans
  Interventions: Drug: Diethylcarbamazine

INTERVENTIONS:
Drug: Diethylcarbamazine — Diethylcarbamazine is a drug administered under an IND held by the CDC. Standard dosing is used.

SUMMARY:
This study will evaluate and treat patients with filarial infections to explore in depth the immunology of the disease, including susceptibility to infection, disease development, and response to treatment. Filarial infections are caused by parasitic worms. The immature worm (larva) is transmitted to a person through a mosquito bite and grows in the human body to 2 to 4 inches in length. Although many of these infections do not produce symptoms, especially in the early stages of infection, others can have serious consequences, including swelling of the limbs or genitalia, allergic-lung problems, skin rash, eye inflammation that can lead to blindness, and heart disease. This protocol does not involve any experimental diagnostic procedures or treatments, and will use only procedures employed in the standard practice of medicine.

Persons between 3 and 100 years of age diagnosed with or suspected of infection with Wuchereria bancrofti, Bugia malayi, Onchocerca volvulus, Loa loa, or other parasitic worms may be eligible for this study.

Participants will have routine tests to determine the specific type of filarial infection. These may include special tests of the lungs, skin or heart, depending on the type of parasite suspected. Patients with skin reactions may have a "punch biopsy" to examine a small piece of affected skin. For this procedure, an area of skin is numbed with an anesthetic and a small circular area, about 1/3-inch in diameter and 1/2-inch thick, is removed using a sharp cookie cutter-type instrument. Some patients may require bronchoalveolar lavage. For this procedure, the mouth and throat are numbed with lidocaine jelly and spray and, if needed, a sedative is given for comfort. A small plastic tube is placed in a vein to give medications. A pencil-thin tube is then passed through the nose or mouth into the lung airways to examine the airways. Salt water is injected through the bronchoscope into the air passage, acting as a rinse. A sample of the fluid is then withdrawn and examined for infection, inflammatory cells and inflammatory chemicals. (Bronchoalveolar lavage is done only if medically necessary and only on patients 21 years or older.) Once the diagnosis is established, standard treatment will be instituted with either diethylcarbamazine or ivermectin, depending on the type of infection.

Additional procedures for research purposes include:

* Extra blood draws to study immune cells and other immune substances. (This is the only research procedure that will be done in - More frequent and extensive follow-up evaluations than usual for routine care. They will include physical examination and blood studies.
* Urine collections at specified periods, possibly including 24-hour collections.
* Skin tests to examine the body s reaction to allergens-common environmental substances, such as cat dander or pollen-that cause an allergic reaction. The test is done in one of two ways: either the skin is lightly scratched and an allergen extract is placed over the just-broken skin, or a very fine needle is used to inject a small amount of allergen under the skin. In both methods, the site is monitored for swelling or hives in the next 48 hours.
* Leukapheresis (only on patients 21 or older ) to collect quantities of white blood cells. Whole blood is collected through a needle in an arm vein, similar to donating blood. The blood circulates through a machine that separates it into its components, and the white cells are removed. The rest of the blood is returned to the body, either through the same needle or through another needle in the other arm.

DETAILED DESCRIPTION:
Patients admitted on this protocol will have, or be suspected of having, one of the filarial infections affecting humans. After routine clinical evaluation they will be studied in depth immunologically, and their blood cells and/or serum will be collected to provide reagents (eg., specific antibodies, T-cell clones, etc.) that will be used in the laboratory to address the broader questions of diagnosis, immunoregulation, pathology and immunoprophylaxis. Careful observations of the patients' clinical and immunologic responses to therapy will be made, as well as long-term follow-up of these changes. It is anticipated both that the patients will receive optimal clinical care for their infections and that the specimens collected from them will prove to be valuable reagents for the laboratory studies of the immunologic responses unique to filarial or other related helminth infections.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age 3-100 years.

Access to a primary medical care provider outside of the NIH.

Ability to give informed consent.

Clinical evidence suggestive of a filarial infection

EXCLUSION CRITERIA:

Although pregnant or nursing women can be enrolled, they will be excluded from receiving treatment while pregnant or breastfeeding

Less than 3 year of age; greater than 100 years of age

Any condition that the investigator feels put the subject at unacceptable risk for participation in the study

Ages: 3 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Males and females having or suspected of having a filarial infections will be enrolled. The participants will either have been native residents of endemic regions where these filarial infections are prevalent or they would have acquired the infection while traveling to such regions.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 1991-03-15 (Actual)

PRIMARY OUTCOMES:
Define the determinants of the susceptibility to filarial infection, the development of filarial disease and the beneficial or adverse response to chemotherapy | 10 years
  Susceptibilities to filarial infection will be determined

SECONDARY OUTCOMES:
To identify clinical and biological markers of successful treatment in filarial-infected individuals | 10 years
  Identification of clinical and biological markers of successful treatments
To characterize the immunoregulatory mechanisms at play in filaria-infected individuals | 10 years
  Characterization of immunoregulatory mechanisms
To create a serum and cell bank for the study of filarial infections of humans both before and at fixed times following definitive treatment. | 10 years
  Cell and serum bank will be maintained.
To understand the natural history of filarial infections in expatriates and other travelers and in immigrant populations | 10 years
  Better understanding of natural history of infections in expatriates and travels

CONTACTS AND LOCATIONS:
Overall Officials: Thomas B Nutman, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Klion AD, Horton J, Nutman TB. Albendazole therapy for loiasis refractory to diethylcarbamazine treatment. Clin Infect Dis. 1999 Sep;29(3):680-2. doi: 10.1086/598654. PMID 10530467
- [Background] Showler AJ, Kubofcik J, Ricciardi A, Nutman TB. Differences in the Clinical and Laboratory Features of Imported Onchocerciasis in Endemic Individuals and Temporary Residents. Am J Trop Med Hyg. 2019 May;100(5):1216-1222. doi: 10.4269/ajtmh.18-0757. PMID 30761981
- [Background] Herrick JA, Metenou S, Makiya MA, Taylar-Williams CA, Law MA, Klion AD, Nutman TB. Eosinophil-associated processes underlie differences in clinical presentation of loiasis between temporary residents and those indigenous to Loa-endemic areas. Clin Infect Dis. 2015 Jan 1;60(1):55-63. doi: 10.1093/cid/ciu723. Epub 2014 Sep 18. PMID 25234520
- [Derived] Bennuru S, Kodua F, Drame PM, Dahlstrom E, Nutman TB. A Novel, Highly Sensitive Nucleic Acid Amplification Test Assay for the Diagnosis of Loiasis and its Use for Detection of Circulating Cell-Free DNA. J Infect Dis. 2023 Oct 3;228(7):936-943. doi: 10.1093/infdis/jiad186. PMID 37243712
- [Derived] Ricciardi A, Nutman TB. IL-10 and Its Related Superfamily Members IL-19 and IL-24 Provide Parallel/Redundant Immune-Modulation in Loa loa Infection. J Infect Dis. 2021 Feb 3;223(2):297-305. doi: 10.1093/infdis/jiaa347. PMID 32561912
- [Derived] Herrick JA, Makiya MA, Holland-Thomas N, Klion AD, Nutman TB. Infection-associated Immune Perturbations Resolve 1 Year Following Treatment for Loa loa. Clin Infect Dis. 2021 Mar 1;72(5):789-796. doi: 10.1093/cid/ciaa137. PMID 32055862
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1988-I-0083.html